CLINICAL TRIAL: NCT02449525
Title: Extracorporal Perfusion of Free Flaps in the Head and Neck
Brief Title: Extracorporeal Perfusion of Microvascular Free Flaps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, thomas.muecke, ECP Study, Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKG-ECP
Record Dates: First submitted 2015-05-11; First posted 2015-05-20 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Perfusion; Complication of Perfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- perfusion of flaps by a bypass system (Experimental): Support of perfusion of microvascular free flaps until ingrowth of vessels from the wound bed has taken place. The System works with a pressure controlled bypass to ensure low grade perfusion.
  Interventions: Procedure: Perfusion of flaps by a special bypass system

INTERVENTIONS:
Procedure: Perfusion of flaps by a special bypass system — Free flaps are perfused via a special bypass perfused by a new technique supported by a intermittent perfusion support system.

SUMMARY:
The perfusion of microvascular free flaps is inevitable for completion of reconstruction in the head and neck area. In some patients microvascular anastomosis is impossible because of arteriosclerotic changes, different oncological interventions, and consecutive vessel depletion at the neck. The aim of the project is to establish an innovative system for extracorporeal perfusion of microvascular free flaps after ingrowth of new vessels from the wound bed have taken place. Afterwards, no further perfusion of the vascular pedicle is required for free flaps to survive and provide functional and aesthetic reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Vessel depleted neck
* defect in the head and neck area

Exclusion Criteria:

* active oncological disease
* vessels suitable for microvascular anastomosis and reconstruction

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-06; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Perfusion of Free Flap from wound bed | Two Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Klaus-Dietrich Wolff, Univ.-Prof., Study Director — Technical University of Munich
Locations (1):
- Department of Oral and Maxillofacial Surgery, Technische Universität München, Munich, Germany

REFERENCES:
- [Derived] Fichter AM, Ritschl LM, Rau A, Schwarzer C, von Bomhard A, Wagenpfeil S, Wolff KD, Mucke T. Free flap rescue using an extracorporeal perfusion device. J Craniomaxillofac Surg. 2016 Dec;44(12):1889-1895. doi: 10.1016/j.jcms.2016.09.010. Epub 2016 Sep 23. PMID 27756552
- [Derived] Wolff KD, Mucke T, von Bomhard A, Ritschl LM, Schneider J, Humbs M, Fichter AM. Free flap transplantation using an extracorporeal perfusion device: First three cases. J Craniomaxillofac Surg. 2016 Feb;44(2):148-54. doi: 10.1016/j.jcms.2015.11.007. Epub 2015 Dec 1. PMID 26752222